CLINICAL TRIAL: NCT02010918
Title: A Phase III, Multicenter, Randomized, Parallel, Open Label and Comparative Study to Evaluate the Efficacy of 500 mg Glucosamine Sulfate (GS) / 400 mg Chondroitin Sulfate (CS)Capsules and 1500 mg GS / 1200 mg CS Sachet Compared With Cosamin DS® Capsule in Treatment of Knee Osteoarthritis..
Brief Title: Efficacy and Safety of Glucosamine Sulfate and Chondroitin Sulfate Combination in Treatment of Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACH-ART-03(01/08)
Record Dates: First submitted 2013-07-19; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis;; Glucosamine;; Chondroitin.
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Glucosamine; Chondroitin Sulfates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- glucosamine sulfate /chondroitin sulfate capsule (Experimental): 500 mg glucosamine sulfate + 400 mg chondroitin sulfate - capsules; One capsule, three times daily.
  Interventions: Drug: glucosamine sulfate /chondroitin sulfate - capsules
- glucosamine sulfate /chondroitin sulfate - sachet (Experimental): 1500 mg glucosamine sulfate / 1200 mg chondroitin sulfate - sachet; One sachet preparation, once daily.
  Interventions: Drug: glucosamine sulfate /chondroitin sulfate - sachet
- Cosamin DS® (Active Comparator): 500 mg glucosamine hydrochloride + 400 mg chondroitin sulfate - Capsules; One capsule, three times daily.
  Interventions: Drug: Cosamin DS®

INTERVENTIONS:
Drug: glucosamine sulfate /chondroitin sulfate - capsules — 500 mg glucosamine sulfate + 400 mg chondroitin sulfate - capsules; One capsule, three times daily.
  Arms: glucosamine sulfate /chondroitin sulfate capsule
Drug: glucosamine sulfate /chondroitin sulfate - sachet — 1500 mg glucosamine sulfate / 1200 mg chondroitin sulfate - sachet; One sachet preparation, once daily.
  Arms: glucosamine sulfate /chondroitin sulfate - sachet
Drug: Cosamin DS® — 500 mg glucosamine hydrochloride + 400 mg chondroitin sulfate - Capsules; One capsule, three times daily.
  Arms: Cosamin DS®

SUMMARY:
The purpose of this study is to determine whether 500 mg Glucosamine Sulfate / 400 mg Chondroitin Sulfate Capsules and 1500 mg Glucosamine Sulfate / 1200 mg Chondroitin Sulfate Sachet is effective and safe compared Cosamin DS ® Capsule in Treatment of Knee Osteoarthritis.

DETAILED DESCRIPTION:
The Groups receive treatment for 16 weeks. The study is realized in 16 sites in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, older than 40 years of age, with knee osteoarthritis, based on clinical and radiological criteria (Kellgren-Lawrence grade 2 - 3), as specified:

  1. Pain on movement of the affected knee for more than 15 days in the previous month with at least partial relief at rest;
  2. Presence of osteophytes at least 1 mm in radiological imaging;
* Knee osteoarthritis symptoms for at least six months prior to randomization.

Exclusion Criteria:

* Concomitant arthropathy that may confuse or interfere with assessing the efficacy or pain;
* Patellar disease isolated, with primary symptoms of pain in the anterior knee, in the absence of radiological findings already described;
* History of significant injury on collateral ligament, or anterior cruciate, or meniscus of the joint studied, with surgery, or immobilization for at least 3 weeks;
* Arthroscopy of the affected knee in last 6 months;
* Serum creatinine ≥ 1.8 mg/dL;
* Diagnosis of diabetes mellitus;
* Presence of any serious disease that could compromise the study, at the investigator discretion;
* History of adverse event or allergy to acetaminophen, glucosamine sulfate or chondroitin sulfate;
* Inability to understand and report the study questionnaire and the Visual Analogic Scale;
* Inability to understand and consent to participate in this clinical study, expressed by signing the Informed Consent (IC);
* Woman in pregnancy.
* If female of childbearing potential, has a negative urine pregnancy test at Visit 0 and do not use, or do not agree to use, for the duration of the study, a medically acceptable form of contraception as determined by the investigator;
* Alcohol intake ( > 3 doses/day);
* Oral or intramuscular corticosteroids four weeks prior to study entry;
* Intra-articular injections with corticosteroids, into the studied knee, within the past three months;
* Intra-articular injections in any other joint within the past four weeks;
* NSAID users that don´t respect the washout period. Low-dose aspirin (325 mg or less, once daily) is allowed for cardio-protective benefit;
* Intra-articular injections of hyaluronic acid within the past 12 months;
* Use of topical analgesic in the joint studied or any other oral analgesic (with the exception of acetaminophen and other NSAID) two weeks prior to randomization;
* Implementation of any other medical treatment for osteoarthritis one month prior to study entry;
* Participation in last one year of clinical protocols, unless it can be direct benefit to patient;
* Use of glucosamine and/or chondroitin sulfate three and six months prior the study entry, respectively;
* Initiation of physical therapy two months prior to the study period;
* Use of tetracycline and oral anticoagulants;
* Use of vitamin D in doses in doses above the recommended;
* Patients in alternative therapies;
* Allergy to sulfonamides;
* Presence of psychiatric disorders that could compromise the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 922 (Actual)
Dates: Start 2009-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain intensity in the affected knee and variation of Lequesne's index and VAS at week 16 . | BASELINE, week 16

SECONDARY OUTCOMES:
Percentage of Participants with any Decrease in Pain Visual Analogue Scale (VAS) | baseline, week 16

OTHER OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | baseline, week 16

CONTACTS AND LOCATIONS:
Overall Officials: José R Provenza, MD, Principal Investigator — Pontifícia Universidade Católica de Campinas, São Paulo, Brazil
Locations (1):
- Serviço de reumatologia do hospital e maternidade celso pierro da PUC-Campinas, Campinas, São Paulo, Brazil